CLINICAL TRIAL: NCT04281095
Title: A Phase I/II Randomized, Double Blind, Active-controlled, Single Center Clinical Trial for Evaluation of Safety and Efficacy of ATGC-110, An Intramuscularly Administered Clostridium Botulinum Neurotoxin Type A, in Adult Patients With Moderate to Severe Glabellar Frown Lines
Brief Title: A Comparative Study of Botulinum Neurotoxin Type A in Treatment of Moderate to Severe Glabellar Frown Lines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ATGC Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBAP-PLN-001
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin type A(ATGC-110) (Experimental)
  Interventions: Drug: Botulinum toxin type A
- Botulinum toxin type A (Active Comparator)
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Total of 20U/0.5mL is intramuscularly administered to five points of the glabellar region, 4U/0.1mL each

SUMMARY:
Efficacy and safety of the investigational product, ATGC-110, was evaluated in comparison with Botox for a total of 12 weeks after the administration in treatment of glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 19 to 65 years
* Subjects assigned a glabellar line severity grade of 2 or greater (moderate) at maximum frown assessed by the Investigator
* Subjects who provide written consent to voluntarily participate in the study after receiving and understanding a detailed explanation of the study

Exclusion Criteria:

* Subjects with diseases that may affect neuromuscular function, such as Myasthenia gravis, Lambert-Eaton syndrome, Amyotrophic lateral sclerosis, or motor neuropathy
* Subjects with the history of eyelid paralysis or ptosis
* Subjects with significant facial asymmetry
* Individuals whose glabellar lines cannot be satisfactorily improved with physical methods since lines are not flattened even using hands
* Subjects who have received medication that inhibits neuromuscular function within the 4 weeks prior to screening such as muscle relaxants, anticholinergics, benzodiazepines and similar drugs, benzamides, tetracycline antibiotics, lincomycin antibiotics, and aminoglycoside antibiotics
* Subjects taking anticoagulants or antiplatelet agents (Use of low-dose aspirin (325 mg/day or less) to prevent blood clotting is allowed)
* Subjects who have received aspirin or NSAIDs within 7 days prior to administration of the IP.
* Subjects with skin abnormalities such as infection at the injection site, dermatopathy, or scars.
* Subjects with the history of treatment of the glabellar region (including the forehead) such as face lifting, permanent implants, or fillers
* Subjects who have received other procedures that may affect the assessment of the glabellar or forehead lines during the following periods:

  * Within 6 months of screening: facial plastic surgery such as tissue augmentation, brow lift, or dermal resurfacing.
  * Within 6 months of screening: injection of dermal fillers with hyaluronic acid as the main ingredient.
  * Within 12 months of screening: injection of dermal fillers with ingredients other than hyaluronic acid as the main ingredient.
* Individuals planning a facial cosmetic procedure (skin fillers, photorejuvenation, chemical/mechanical peeling, etc.) during the study period.
* Individuals who have received a botulinum toxin preparation within 5 months prior to screening or those who are expected to receive a botulinum toxin preparation for any other purpose than the indication of this study (glabellar lines).
* Subjects with the history of excessive alcohol consumption or drug addiction
* Individuals with an anxiety disorder or other significant psychiatric disorders (e.g., depression), which, in the Investigator's opinion, may affect study participation or objective assessment of efficacy outcomes
* Individuals who answered "yes" to any of the questions on the Columbia University Suicide Severity Rating Scale (C-SSRS) regarding a case within the past 12 months at the screening
* Female subjects of childbearing age who do not agree to practice contraception using medically allowed contraceptive methods during the study period (hormonal contraception, IUD (intrauterine device) or IUS (intrauterine system), tubal ligation, dual protection (using a combination of male condom, female condom, cervical cap, contraceptive diaphragm, or contraceptive sponge)
* Pregnant or lactating women
* Subjects who are allergic or sensitive to the IP or its components
* Individuals with concomitant illnesses that make them unsuitable for participation in the study by the Investigator such as malignant tumors, immunodeficiency (immune deficiency), kidney disease, liver disease, or lung disease
* Individuals who have participated in other clinical trials within 3 months prior to participating in this study and have received an IP or medical device during the previous clinical studies
* Individuals who are not eligible for this study for any reason as per the Investigator's discretion

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment | 0 and 4 weeks after the administration
  Changes in the glabellar line severity at maximum frown from baseline to 4 weeks after the IP administration were evaluated by investigator

SECONDARY OUTCOMES:
Glabellar line improvement rate at maximum frown confirmed by investigator's live assessment | 0, 8, 12 weeks after the administration
  Changes in the glabellar line severity at maximum frown from baseline to 8 and 12 weeks after the IP administration were evaluated by investigator
Glabellar line improvement rate at rest confirmed by investigator's live assessment | 0, 4, 8, 12 weeks after the administration
  Changes in the glabellar line severity at rest from baseline to 4, 8 and 12 weeks after the IP administration were evaluated by investigator
Glabellar line improvement rate at rest confirmed by subject's assessment | 0, 4, 8, 12 weeks after the administration
  Changes in the glabellar line severity at rest from baseline to 4, 8 and 12 weeks after the IP administration were evaluated by subjects
Subject satisfaction rate | 0, 4, 8, 12 weeks after the administration
  Subjects fill out the satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nowon Eulji Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No